CLINICAL TRIAL: NCT05150808
Title: WHO Phase III Evaluation of Vectron T500 (Broflanilide 50WP) for IRS in Tanzania
Brief Title: Vectron T500 (Broflanilide 50WP) for IRS in Tanzania Tanzania
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government); Kilimanjaro Christian Medical Centre, Tanzania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ph3 Vectron Tz; ITDCZI93 (Other Grant/Funding Number: IVCC)
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Malaria,Falciparum
Keywords: vector control; insecticide; indoor residual spraying of mosquitoes
MeSH Terms: conditions — Malaria, Falciparum | interventions — 3-benzamido-N-(4-(perfluoropropan-2-yl)phenyl)benzamide

STUDY DESIGN:
Intervention Model Description: Cluster Randomised Trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention IRS (Active Comparator): Intervention IRS insecticide will be sprayed on the walls and ceilings of 8 clusters
  Interventions: Other: IRS insecticide: Vectron T500
- Control IRS (Active Comparator): WHO approved IRS insecticide will be sprayed on the walls and ceilings of 8 clusters
  Interventions: Other: IRS insecticide: Vectron T500

INTERVENTIONS:
Other: IRS insecticide: Vectron T500 — public health insecticide
  Other Names: broflanilide

SUMMARY:
Malaria is a major public health problem in Africa. An important way to control the disease is by Indoor Residual Spraying of insecticide in houses. Insecticide resistance has become a major problem. This trial will evaluate a novel insecticide against those insecticide resistant mosquito vectors in Tanzania E Africa.

DETAILED DESCRIPTION:
Background: Indoor residual spraying (IRS) is one of the major methods of malaria vector control across sub-Saharan Africa, responsible for reducing malaria incidence by 10% since 2000. However, effective vector control is increasingly threatened by the rapid spread of insecticide resistance. Consequently, there have been investments in the development of new insecticides for IRS that possess novel modes of action with long residual activity, low mammalian and environmental toxicity and minimal cross-resistance. VECTRONTM T500, a new IRS insecticide containing the active ingredient broflanilide 50% WP, has been shown to be efficacious against both pyrethroid-susceptible and -resistant vector strains on mud and concrete substrates in phase II experimental hut trials in Tanzania.

Method: A two-arm non-inferiority cluster randomized controlled trial will be conducted in Muheza District, Tanga Region, Tanzania. VECTRONTM T500 will be compared to the IRS formulation Fludora® Fusion (active ingredients: clothianidin 50% WP + deltamethrin 6.25% WP). The predominant malaria vectors in the study area are pyrethroid-resistant Anopheles gambiae s.s., An. arabiensis and An. funestus s.s. Sixteen selected clusters of 75-200 households in each cluster will be pair-matched on baseline vector densities and allocated to reference and intervention arms. Consenting households in the intervention arm will be sprayed with VECTRONTM T500 and those in the reference arm will receive Fludora® Fusion. Monthly CDC light traps will collect mosquitoes to determine vector density, indoor biting, sporozoite and entomological inoculation rates (EIR). Phenotypic resistance to IRS active ingredients will be assessed using CDC bottle bioassays. Molecular and metabolic resistance mechanisms will be characterised among Anopheles field populations from both trial arms. Residual efficacy of both brands of insecticide will be monitored for 12 months post-spraying. A semi-structured questionnaire and focus group discussions will explore social and cultural factors that influence acceptability, perceived adverse effects and benefits of IRS.

Discussion: This protocol describes a phase III non-inferiority evaluation of a novel IRS product to reduce the density and EIR of pyrethroid-resistant Anopheles vectors. If VECTRONTM T500 proves non-inferior to Fludora® Fusion, it may be considered as an additional vector control product for malaria prevention and insecticide resistance management schemes.

ELIGIBILITY:
Inclusion Criteria:

All households who consent to IRS malaria control

Exclusion Criteria:

none

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12500 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Vector density | 12-15 months
  Reduction in vector population density
Sporozoite rate | 12-15 months
  Reduction in sporozoite rate
Entomological inoculation rate EIR | 12-15 months
  Reduction in EIR

CONTACTS AND LOCATIONS:
Locations (2):
- National Institute of Medical Research, Muheza, Tanzania
- London School of Hygiene & Tropical Medicine, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mbewe NJ, Tungu PK, Messenger LA, Bradley J, Mangesho PE, Shirima B, Moshi O, Shayo MF, Seif M, Portwood NM, Snetselaar J, Azizi S, Magogo F, Mabenga P, Sudi W, Mlay G, Kirby MJ, Mosha FW, Kisinza W, Matowo J, Small G, Rowland MW. A noninferiority cluster randomised evaluation of a broflanilide indoor residual spraying insecticide, VECTRON T500, for malaria vector control in Tanzania. Sci Rep. 2025 Apr 29;15(1):15013. doi: 10.1038/s41598-025-99809-9. PMID 40301570
- [Derived] Tungu PK, Rowland MW, Messenger LA, Small GJ, Bradley J, Snetselaar J, Kirby MJ, Mbewe NJ. Large-scale (Phase III) evaluation of broflanilide 50WP (VECTRON T500) for indoor residual spraying for malaria vector control in Northeast Tanzania: study protocol for a two-arm, non-inferiority, cluster-randomised community trial. BMC Infect Dis. 2022 Feb 21;22(1):171. doi: 10.1186/s12879-022-07138-3. PMID 35189830